CLINICAL TRIAL: NCT00816764
Title: A Phase 1, Open-label, Multi-center, Dose Escalation Study of the Safety and Pharmacokinetics of AGS-8M4 Given as Monotherapy in Subjects With Advanced Ovarian Cancer
Brief Title: A Phase 1 Study of the Safety and Pharmacokinetics of AGS-8M4 in Subjects With Advanced Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Agensys, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008001
Record Dates: First submitted 2009-01-01; First posted 2009-01-05 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2010-11

CONDITIONS: Carcinoma; Ovarian Cancer; Ovarian Diseases; Ovarian Neoplasms
Keywords: clinical trial, phase 1; carcinoma; pharmacokinetics; safety; ovarian
MeSH Terms: conditions — Carcinoma; Ovarian Neoplasms; Ovarian Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1. AGS-8M4 Dose 1 (Experimental)
  Interventions: Biological: AGS-8M4
- 2. AGS-8M4 Dose 2 (Experimental)
  Interventions: Biological: AGS-8M4
- 3. AGS-8M4 Dose 3 (Experimental)
  Interventions: Biological: AGS-8M4
- 4. AGS-8M4 Dose 4 (Experimental)
  Interventions: Biological: AGS-8M4

INTERVENTIONS:
Biological: AGS-8M4 — IV Infusion

SUMMARY:
This is the first in human study of AGS-8M4 given every 2 weeks to subjects with advanced ovarian cancer. AGS-8M4 will be administered as an IV infusion until the disease worsens.

DETAILED DESCRIPTION:
All Subjects will receive AGS-8M4 treatment. Subjects will be enrolled sequentially into 1 of the 4 planned dose cohorts according to a standard dose escalation study design. A disease assessment will be performed at study week 9 (+/- 3 days). The assessment will be based on clinical signs and symptoms, changes in radiographic images, and changes in CA-125 levels. Subjects without evidence of disease progression may continue to receive AGS-8M4 during the extended treatment period at the dose and schedule of their assigned cohort until disease progression intolerability of AGS-8M4 or consent withdrawal. For subjects that continue dosing, disease assessments will be performed every 8 weeks during the extended treatment period. A safety follow-up visit will occur 4 weeks after the last infusion of AGS-8M4.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with recurrent disease or histologically or cytologically confirmed Stage III/IV diagnosis of epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal carcinoma
* Subjects must have received at least one prior platinum containing regimen and one of the following: persistent disease (either stable disease, partial response or nonmeasureable disease after first line therapy) or progressive disease at anytime

Exclusion Criteria:

* No epithelial ovarian tumors of low malignant potential
* Active infection requiring treatment with systemic anti-infectives within 72 hours of screening
* Use of any investigational drug within 30 days prior to screening or 5 half-lives of the prior investigational drug (whichever is longer)
* Prior monoclonal antibody therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Throughout the treatment
Assessment of PK variables | Weeks 1-3, week 5, week 7 week 11, every 2 weeks during extension period, 2 and 3 months after last dose

SECONDARY OUTCOMES:
Incidence of anti-AGS-8M4 antibody formation | Week 1, week 7, week 11, week 15 (extension only), 2 and 3 months after last dose
Changes in tumor status per RECIST | Week 9, and every 8 weeks during the extended treatment period
Changes in CA-125 levels | Week 9, and every 8 weeks during the extended treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Agensys, Inc.
Locations (2):
- United States (2):
  - Baltimore, Maryland
  - New York, New York